CLINICAL TRIAL: NCT03710785
Title: Analysis of Abnormal Muscle Activities on Forward Neck Posture Syndrome Patients and Effect of Neck Extension Exercise Using 8 Channel Surface Electromyography
Brief Title: Effect of Neck Extension Exercise Using 8 Channel Surface Electromyography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ju Seok Ryu, associate professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: B-1709/421-005
Record Dates: First submitted 2018-10-07; First posted 2018-10-18 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Neck Syndrome
Keywords: 8 Channel Surface Electromyography; Forward Neck Posture Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- forward neck posture syndrome patients (Experimental): Patients diagnosed with forward neck posture syndrome in cervical plain X-ray have a cervical spine extension exercise for 4 weeks
  Interventions: Behavioral: cervical spine extension exercise

INTERVENTIONS:
Behavioral: cervical spine extension exercise — cervical spine extension exercise for 4 weeks

SUMMARY:
Analysis of Abnormal Muscle Activities on Forward Neck Posture Syndrome Patients and Effect of Neck Extension Exercise Using 8 Channel Surface Electromyography

DETAILED DESCRIPTION:
In this study, the investigators investigate the muscle contraction according to posture change in patients with forward neck posture syndrome which was not revealed by 8 channel surface electromyography and provide accurate evaluation of forward neck posture syndrome in comparison with normal group and to be used as basic research data for the development of 8 channel electric stimulation therapy device.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults over the age of 20 who do not have any underlying disease that does not appeal to forward neck posture syndrome 2) Among adults who complained of chronic pain over three months, patients aged 20 years and over who were diagnosed with forward neck posture syndrome in a simple x-ray of the lumbar spine

Exclusion Criteria:

* Patients with severe neurological disorders (procedural hypertrophy), previous cervical surgery, impaired eye diseases, spinal deformations, rehabilitation for strengthening spinal muscles within the last three months and pregnant women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-09-18 (Actual)

PRIMARY OUTCOMES:
Change from 8 Channel Surface Electromyography at 4 weeks | when patient enrolled and after 4 weeks
  measure the area and extent of muscle activation around the cervical vertebrae according to posture

SECONDARY OUTCOMES:
Change the angle of cervical vertebrae from plain x-ray at 8 weeks | when patient enrolled and after 8 weeks
  measure the angle of cervical vertebrae

CONTACTS AND LOCATIONS:
Overall Officials: Jusuk Ryu, M.D. PhD, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Lim J, Lee D, Kim S, Lee S, Ryu JS. Analysis of abnormal muscle activities in patients with loss of cervical lordosis: a cross-sectional study. BMC Musculoskelet Disord. 2023 Aug 22;24(1):666. doi: 10.1186/s12891-023-06782-3. PMID 37608321